CLINICAL TRIAL: NCT01033838
Title: Conventional Laparoscopic-assisted Rectosigmoid Resection Versus Laparoscopic Rectosigmoid Resection With Intracorporeal Anastomosis and Transrectal Specimen Retrieval
Brief Title: Randomized Trial Comparing Laparoscopic-assisted Rectosigmoid Resection Versus Laparoscopic Rectosigmoid Resection With Transrectal Specimen Retrieval
Acronym: LATA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Prof. Dr. A. D'Hoore, Universitaire Ziekenhuizen Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S51801-B32220097328
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Symptomatic Recurrent Diverticular Disease; Benign Adenomatous Sigmoidal Polyp, Requiring Surgery; Early Non-transmural Sigmoidtumor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- laparoscopic-assisted rectosigmoid resection (Active Comparator)
  Interventions: Procedure: rectosigmoid resection
- laparoscopic rectosigmoid resection and transrectal retrieval (Experimental)
  Interventions: Procedure: rectosigmoid resection

INTERVENTIONS:
Procedure: rectosigmoid resection

SUMMARY:
Laparoscopic anterior resection is a standardized procedure requiring a small muscle split incision to retrieve the specimen and to fashion the proximal part of the double stapled anastomosis. Most patients can be included within a standardized perioperative care program called Enhanced Recovery After Surgery (ERAS). A new evolution as a primary step towards a complete Natural Orifice Translumenal Endoscopic Surgery (NOTES)-procedure is a hybrid approach (transrectal and laparoscopic). The dissection is performed laparoscopically but the specimen is retrieved within an endobag through the rectum. The anastomosis is created intracorporeally using a triple stapled technique. There are no trials available in the literature concerning these 2 techniques. Therefore this study will be undertaken to establish the role of the 2 surgical procedures and to compare them after short-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Symptomatic recurrent diverticular disease
* Benign adenomatous polyp, requiring surgery
* Early non-transmural sigmoidtumor
* Signed written informed consent, approved by ethical committee

Exclusion Criteria:

* Patients unsuitable for laparoscopy
* Pregnancy
* ASA >III
* Coagulation disorders
* Anti-coagulants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in analgetic need

SECONDARY OUTCOMES:
reduction in hospital stay within an ERAS-program
effect on the inflammatory response
effect on anal continence
procedural cost assessment (incorporating operative time)
overall cost assessment

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Wolthuis AM, Fieuws S, Van Den Bosch A, de Buck van Overstraeten A, D'Hoore A. Randomized clinical trial of laparoscopic colectomy with or without natural-orifice specimen extraction. Br J Surg. 2015 May;102(6):630-7. doi: 10.1002/bjs.9757. Epub 2015 Mar 12. PMID 25764376